CLINICAL TRIAL: NCT01501357
Title: Effectiveness of Toothbrushing Techniques in Plaque Removal and Caries Lesion Control in Erupting Primary Permanent Molars - Randomized Clinical Trial Abbreviated Over 24 Months
Brief Title: Effectiveness of Toothbrushing Techniques in Plaque Removal and Caries Lesion Control
Acronym: toothbrushing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mariana Minatel Braga, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Caries
Keywords: caries; primary molars; plaque; toothbrushing
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multilevel filaments toothbrush (Experimental): Children will brush with anteroposterior toothbrushing and a modified toothbrush (multilevel filaments)
  Interventions: Behavioral: modified toothbrush with multilevel filaments
- cross toothbrushing (Active Comparator): Children will brush with cross toothbrushing.
  Interventions: Behavioral: cross toothbrushing

INTERVENTIONS:
Behavioral: modified toothbrush with multilevel filaments — After the allocation of patients in this group they were instructed to brush their first molars erupt with the brushing technique anteroposterior.
  Other Names: stages, oral b
  Arms: multilevel filaments toothbrush
Behavioral: cross toothbrushing — Children allocated to the group multi-bristled brush will be modified compared to the results of the group cross toothbrushing technique
  Other Names: buccal-lingual technique
  Arms: cross toothbrushing

SUMMARY:
The aim of the study is to evaluate the effectiveness of cross-toothbrushing technique compared with anteroposterior and biofilm removal and control of caries lesions in first permanent molars.

DETAILED DESCRIPTION:
220 children between 5-7 years with at least one permanent molar erupting will be selected, with a maximum score of ICDAS 3. These children will be randomly allocated into two groups according to the technique adopted. The teeth will be evaluated by ICDAS, laser fluorescence (DIAGNOdent), QLF and subtraction radiography at baseline and after 15 days, 3, 6, 9,12,18,24 months.

ELIGIBILITY:
Inclusion Criteria:

* erupting primary permanent molar

Exclusion Criteria:

* caries ( ICDAS 4,5 and 6),
* enamel defects,
* sealant,
* restoration

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
dental caries | 24 months

SECONDARY OUTCOMES:
dental plaque | 24 months
  Dental plaque accumulation after short and long term analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mariana M Braga, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, Brazil